CLINICAL TRIAL: NCT05341661
Title: A Prospective, Randomized, Controlled, Blinded Study to Assess the Safety and Efficacy of the Butterfly Medical Prostatic Retraction Device in BPH Patients
Brief Title: Butterfly Pivotal Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butterfly Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-BM14-001
Record Dates: First submitted 2021-12-20; First posted 2022-04-22 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: BPH (Benign Prostatic Hyperplasia); Lower Urinary Tract Symptoms (LUTS)
Keywords: BPH, LUTS
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Active (Active Comparator): The active arm patients undergo the Butterfly device procedure.
  Interventions: Device: Butterfly Prostatic Retraction Device
- Sham Comparator (Sham Comparator): The sham control arm patients undergo a rigid cystoscopy procedure.
  Interventions: Device: Butterfly Prostatic Retraction Device
- Cross over (Other): Sham arm patient is allowed to crossover and undergo the Butterfly procedure
  Interventions: Device: Butterfly Prostatic Retraction Device

INTERVENTIONS:
Device: Butterfly Prostatic Retraction Device — Implantation of the Butterfly device

SUMMARY:
A prospective, multicenter, blind randomized (2:1) controlled study comparing the International Prostate Symptom Score (IPSS) of the Active arm to the IPSS of the control arm at the 3 months follow-up and active arm IPSS score change from time zero to 12 months. Patients in the active arm undergo Butterfly device treatment. Patients in the control arm undergo a sham rigid cystoscopy procedure

ELIGIBILITY:
Inclusion Criteria:

1. Male patient age 50 and up
2. Willing and able to sign informed consent
3. Willing and able to comply with all study assessments
4. Prostate length of 25mm-45mm (from apex of the prostate to the beginning of the bladder neck).
5. Prostate volume 30-90 ml
6. Symptomatic BPH: IPSS ≥ 13; ≥ 1 in the IPSS voiding to sub-score ratio (IPSS-V/S)

Exclusion Criteria:

1. Known sensitivity to Nickel.
2. Current urinary retention
3. Urinary stress incontinence (sphincter)
4. Biopsy of the prostate within the last 6 weeks
5. Baseline PSA > 10 ng/mL or confirmed or suspected prostate cancer. Patients with a PSA level above 2.5 ng/mL, in which free PSA is < 25% of total PSA in whom cancer was not ruled out by biopsy.
6. Chronic prostatitis, recurrent prostatitis, chronic pelvic pain syndrome (CPPS), or painful bladder syndrome within the past 12 months
7. Obstructing intraprostatic median lobe (e.g., more than 10mm intravesical prostatic protrusion).
8. Urethral stricture, meatal stenosis, or bladder neck stricture - either current or recurrent.
9. Anatomical anomalies that will not accommodate the retractor, as determined by cystoscopy (e.g., prostatic urethral length to height geometry, absence of bladder neck)
10. Prior surgery or minimal invasive procedure of prostate (brachytherapy and PAE patients are not excluded if they show significant obstruction in urodynamic test and cystoscopy shows no significant fibrosis).
11. Currently active bladder tumor or intravesical instillation.
12. History of other diseases causing voiding dysfunction including urinary retention (e.g., uncontrolled diabetes, diagnosis of neurogenic or atonic bladder, Parkinson's disease, multiple sclerosis, etc.).
13. Suspected Neurogenic or atonic urinary bladder.
14. Suspected Polyuria/Nocturnal Polyuria.
15. Suspected overactive bladder
16. High bladder neck with the absence of lateral lobe encroachment indicating a high likelihood of primary bladder neck obstruction as determined by the Investigator
17. Urethral pathology: diverticula, strictures, tumors, fistula.
18. Acute clinically Significant urinary tract infection.
19. Uncontrolled bleeding disorders.
20. Active stone disease (urinary stone increase in size during the last 3 months/ stone passage during the last 3 months/ presence of cystolithiasis)
21. Taking 5 alpha reductase inhibitors within 6 months of baseline evaluation
22. Taking one of the following within 2 weeks of baseline evaluation:

    1. alpha-blockers,
    2. imipramine,
    3. anticholinergics,
    4. Phosphodiesterase-5 Enzyme Inhibitors (Tadalafil) in doses for BPH,
    5. Beta-3 adrenergic receptor agonist (Mirabegron),
23. Taking androgens, unless eugonadal state for at least 2 months or greater as documented by the Investigator
24. Taking Gonadotrophin releasing hormone analogues within 12 months of baseline evaluation
25. Taking one of the following within 24 hours of pre-treatment (baseline) evaluation:

    phenylephrine, or, pseudoephedrine,
26. One of the following baseline test results, taken from a single uroflowmetry reading:

    * Urinary volume void ≤ 125mL (pre-bladder urinary volume of ≥ 150 mL required),
    * Peak urinary flow rate (Qmax) of ≤ 5 ml/second and > 15 mL/second,
    * Post- void residual volume (PVR) > 250 mL
27. Inmates, patient with physical, psychological (such as developmentally delayed adults), or medical impairment that might prevent study completion or would confound study results (including patient questionnaires) in the judgment of the Investigator
28. Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.

Ages: 50 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male age 50 years old and up, suffering from LUTS due to BPH
Enrollment: 245 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to month 3 in International Prostate Symptom Score (IPSS) Score. | 3 month
  Analysis will compare the active and control study arms IPSS
Change in active arm International Prostate Symptom Score (IPSS) from baseline to 12 months | 12 month
  Analysis will assess the IPSS percent change for the active arm compared to a baseline score

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Paz, MD, Study Director — Medical director
Locations (3):
- United States (3):
  - Manhattan Medical Research, New York, New York
  - Northwell Health, Syosset, New York
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No